CLINICAL TRIAL: NCT00820105
Title: A Phase 2B, Randomised, Double-blind, Placebo-controlled, Parallel Group, Dose-ranging, Multicentre Study to Investigate the Efficacy, Safety and Tolerability of the mGluR5 Negative Allosteric Modulator ADX10059 for the Prevention of Migraine
Brief Title: ADX10059 Migraine Prevention Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Incidence of abnormalities of liver function tests is higher than expected in this population.
Sponsor: Addex Pharma S.A. (Industry)
Responsible Party: Study Director, Addex Pharma SA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ADX10059-206; 2008-005481-30
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Migraine
Keywords: Migraine; Aura; Migraine headache
MeSH Terms: conditions — Migraine Disorders; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ADX10059 25 mg (Experimental): Weeks 1-2: once daily Weeks 3-12: twice daily
  Interventions: Drug: ADX10059
- ADX10059 50 mg (Experimental): Weeks 1-2: once daily Weeks 3-12: twice daily
  Interventions: Drug: ADX10059
- ADX10059 100 mg (Experimental): Weeks 1-2: once daily Weeks 3-12: twice daily
  Interventions: Drug: ADX10059
- ADX10059 Matching Placebo (Placebo Comparator): Weeks 1-2: once daily Weeks 3-12: twice daily
  Interventions: Drug: ADX10059 Matching Placebo

INTERVENTIONS:
Drug: ADX10059 — oral administration
  Arms: ADX10059 25 mg
Drug: ADX10059 — Oral administration
  Arms: ADX10059 50 mg
Drug: ADX10059 — Oral administration
  Arms: ADX10059 100 mg
Drug: ADX10059 Matching Placebo — Oral administration
  Arms: ADX10059 Matching Placebo

SUMMARY:
Evaluation of ADX10059 to prevent migraine attacks

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 to 65 years
* History of migraine
* Aged ≤ 50 years at onset of migraine history

Exclusion Criteria:

* Cluster headache or chronic migraine headaches
* Currently uses, or within 3 months of Screening, has used: sodium valproate or topiramate and any other drugs used specifically for migraine prophylaxis, for example beta-blockers, calcium channel blockers, tricyclic antidepressants, selective serotonin reuptake inhibitors
* Unable to distinguish migraine headache from tension and other types of headache
* Current history of psychiatric disorder requiring regular medication
* Known history of alcohol abuse
* Known clinically significant allergy or known hypersensitivity to drugs
* History of a significant medical condition that may affect the safety of the patient or preclude adequate participation in the study
* Pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Number of migraine headache days during weeks 9-12 of the treatment period | 12 weeks

SECONDARY OUTCOMES:
Migraine frequency | 12 weeks
Migraine severity | 12 weeks
Migraine duration | 12 weeks
Occurrence of aura | 12 weeks
Functional impairment severity | 12 weeks
Rescue medication use | 12 weeks
Proportion of responders | 12 weeks
Global assessment of study medication | 12 weeks

CONTACTS AND LOCATIONS:
Locations (31):
- Vienna, Austria
- Belgium (3):
  - Liège, Liège
  - Sint-Truiden, Sint-Truiden
  - Wilrijk, Wilrijk
- France (4):
  - Lille, Lille
  - Nice, Nice
  - Paris, Paris
  - Toulouse, Toulouse
- Germany (18):
  - 06, Berlin
  - Berlin Hellersdorf 11, Berlin
  - Bochum, Bochum
  - Dreseden, Dresden
  - 02, Essen
  - 28, Essen
  - Frankfurt, Frankfurt
  - Freiburg, Freiburg im Breisgau
  - Göppingen, Göppingen
  - Görlitz, Görlitz
  - Hamburg, Hamburg
  - Itzehoe, Itzehoe
  - Leipzig, Leipzig
  - Magdeburg, Magdeburg
  - 05, München
  - 10, München
  - Münster, Münster
  - Wiesbaden, Wiesbaden
- United Kingdom (5):
  - Berkshire, Berkshire
  - Cardiff, Cardiff
  - Liverpool, Liverpool
  - 24, London
  - Manchester, Manchester